CLINICAL TRIAL: NCT02023996
Title: Pilot Trial of PET Imaging With 89Zr-DFO-Trastuzumab in Esophagogastric Cancer
Brief Title: PET Imaging With 89Zr-DFO-Trastuzumab in Esophagogastric Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-165
Record Dates: First submitted 2013-12-18; First posted 2013-12-30 (Estimated); Results first posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2023-06

CONDITIONS: Esophagogastric Cancer
Keywords: HER2 positive; PET Imaging; 89Zr-DFO-trastuzumab; 13-165
MeSH Terms: interventions — zirconium-89-trastuzumab; Positron-Emission Tomography

ARMS (1):
- PET Imaging With 89Zr-DFO-Trastuzumab (Experimental): Patients will receive 5 mCi + 0.5 mCi of 89Zr-DFO-trastuzumab given IV over 5-10 min. Injection of cold trastuzumab will be mixed with 89Zr-DFO-trastuzumab so that total mass is equal to 50 mg [1]. In the first ten patients we wish to obtain normal organ dosimetry, pharmacokinetics & determine optimal imaging time, therefore these patients will undergo imaging at 4 time points post injection, whole body counts & blood draws. Subsequent patients will receive the antibody & will only undergo imaging at a single time point (based on the first 10 patients) & will not have whole body counts or serial bloods for pharmacokinetics. The administration of 89Zr-DFO-trastuzumab to patients undergoing a second study will be identical as for their baseline study. Patients undergoing a second injection will only have one scan that will be performed within 1 day before or 2 days after their optimum imaging time point, determined from their baseline imaging study.
  Interventions: Radiation: 89Zr-DFO-trastuzumab; Device: PET imaging

INTERVENTIONS:
Radiation: 89Zr-DFO-trastuzumab
Device: PET imaging

SUMMARY:
The purpose of the first group (Group 1) was to find the optimal time for taking pictures after injection of 89Zr-DFO-trastuzumab, to see how long it stayed in the blood, and to see how well it was tolerated. From what the investigators have learned from Group 1, patients in Group 2 no longer need serial scans or serial blood draws. This study is based on a cohort expansion. All data is appropriately reported as there is only one study cohort

ELIGIBILITY:
Inclusion Criteria:

* Registered patient at MSKCC
* Age ≥18 years
* Pathologically or cytologically confirmed metastatic or primary esophagogastric cancer HER2 positive status by FISH or IHC as currently being implemented for patients with esophagogastric cancer. HER2 overexpression and/or amplification as determined by immunohistochemistry (3+) or FISH (≥2.0)
* Measurable or evaluable disease, lesions that have not been previously radiated, with clinically indicated imaging evaluation performed within 4 weeks prior to study entry (CT, MRI, FDG PET or bone scan). Patients requiring concurrent radiation treatment are not eligible unless additional lesions that are not being irradiated and are assessable for targeting are present.
* Karnofsky Performance Score ≥ 60
* Ability to understand and willingness to sign informed consent
* Negative pregnancy test, to be performed on female patients of childbearing potential within 1week before administration of radioactive material.
* Life expectancy of at least three (3) months.
* Willingness to use birth control while on study.
* The patients will be asked to consent to provide access to data obtained from molecular analysis that has been done on archived tumor tissue that will be correlated with 89Zr-DFO-trastuzumab imaging results.
* Concurrent therapy will be allowed.

Exclusion Criteria:

* Inability to lie still for the duration of the scanning procedure.
* Patients with known sensitivity or contraindication to any of the component of 89Zr-DFO-trastuzumab (89Zr or Desferroxamine (DFO) or trastuzumab)
* Patients who have received trastuzumab must have at least a washout period for trastuzumab of 14 days, this will not apply to 89Zr-DFO-trastuzumab repeat, post treatment assessment where patients may be receiving trastuzumab.
* HIV positive or active hepatitis.
* History or presence of clinically relevant cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure NYHA classification of 3, unstable angina or poorly controlled arrhythmia. Myocardial infarction within 6 months prior to study entry
* Hematologic

  * Platelets <50K/mcL
  * ANC <1.0 K/mcL
* Hepatic laboratory values

  * Bilirubin >2 x ULN (institutional upper limits of normal), with exception of patients with Gilberts disease. AST/ALT >2.5 x ULN (institutional upper limits of normal); >5 x ULN if liver metastasis
* Renal laboratory values

  * Estimated GFR (eGFR) < 30mL/min/1.73m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neeta Pandit-Taskar, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study is based on a cohort expansion. All data is appropriately reported as there is only one study cohort
Groups:
- PET Imaging With 89Zr-DFO-Trastuzumab: Patients will receive 5 mCi + 0.5 mCi of 89Zr-DFO-trastuzumab given IV over 5-10 min. Injection of cold trastuzumab will be mixed with 89Zr-DFO-trastuzumab so that total mass is equal to 50 mg [1]. In the first ten patients we wish to obtain normal organ dosimetry, pharmacokinetics & determine optimal imaging time, therefore these patients will undergo imaging at 4 time points post injection, whole body counts & blood draws. Subsequent patients will receive the antibody & will only undergo imaging at a single time point (based on the first 10 patients) & will not have whole body counts or serial bloods for pharmacokinetics. The administration of 89Zr-DFO-trastuzumab to patients undergoing a second study will be identical as for their baseline study. Patients undergoing a second injection will only have one scan that will be performed within 1 day before or 2 days after their optimum imaging time point, determined from their baseline imaging study.
  89Zr-DFO-trastuzumab
  PET imaging
Period: Overall Study
Arm/Group | PET Imaging With 89Zr-DFO-Trastuzumab
Started | 42
Completed | 36
Not Completed | 6
Not completed — Protocol Violation | 6

BASELINE CHARACTERISTICS:
Population: This study is based on a cohort expansion. All data is appropriately reported as there is only one study cohort
Arm/Group | PET Imaging With 89Zr-DFO-Trastuzumab
Number analyzed (Participants) | 36
Age, Continuous [Mean (Full Range); unit: years] | 61 [35 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 28
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Safety as Measured by the Number of Participants Who Experienced Toxicity
Description: Participants will be evaluated for toxicity using CTCAE v4.0
Time Frame: 2 years
Population: This study is based on a cohort expansion. All data is appropriately reported as there is only one study cohort
Measure: Count of Participants; unit: Participants
Arm/Group | PET Imaging With 89Zr-DFO-Trastuzumab
Number analyzed (Participants) | 36
Participants
  Participants with toxicity | 2
  Participants without toxicity | 34

2. Primary Outcome: Feasibility of Antibody-imaging
Description: Antibody imaging is considered feasible if 70% of the patients are antibody-imaging positive. Antibody imaging will be considered feasible if 7 or more of the 10 patients in the first cohort are antibody-imaging-positive. We will also require that none of these patients experience severe toxicity attributable to the initial antibody.
Time Frame: 2 years
Population: This study is based on a cohort expansion. All data is appropriately reported as there is only one study cohort
Measure: Count of Participants; unit: Participants
Arm/Group | PET Imaging With 89Zr-DFO-Trastuzumab
Number analyzed (Participants) | 36
Participants
  Participants with >/= 50% tumor load positivity | 24
  Participants with <50% tumor load positivity | 12

3. Secondary Outcome: Biologic Half-time
Description: Samples will be obtained just prior to injection of the 89Zr DFO-trastuzumab tracer this sample will be banked at -80degree C for future testing for Human anti-human antibody/HAHA if altered biodistribution is observed.
Time Frame: Up to 580 hours
Population: This study is based on a cohort expansion. All data is appropriately reported as there is only one study cohort
Measure: Median (Full Range); unit: hours
Arm/Group | PET Imaging With 89Zr-DFO-Trastuzumab
Number analyzed (Participants) | 36
hours | 370 [257 to 578]

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- PET Imaging With 89Zr-DFO-Trastuzumab: Patients will receive 5 mCi + 0.5 mCi of 89Zr-DFO-trastuzumab given IV over 5-10 min. Injection of cold trastuzumab will be mixed with 89Zr-DFO-trastuzumab so that total mass is equal to 50 mg [1]. In the first ten patients we wish to obtain normal organ dosimetry, pharmacokinetics & determine optimal imaging time, therefore these patients will undergo imaging at 4 time points post injection, whole body counts & blood draws. Subsequent patients will receive the antibody & will only undergo imaging at a single time point (based on the first 10 patients) & will not have whole body counts or serial bloods for pharmacokinetics. The administration of 89Zr-DFO-trastuzumab to patients undergoing a second study will be identical as for their baseline study. Patients undergoing a second injection will only have one scan that will be performed within 1 day before or 2 days after their optimum imaging time point, determined from their baseline imaging study.
  This study is based on a cohort expansion. All data is appropriately reported as there is only one study cohort
Arm/Group | PET Imaging With 89Zr-DFO-Trastuzumab
All-Cause Mortality (participants affected / at risk) | 31/36
Serious Adverse Events (participants affected / at risk) | 2/36
Other Adverse Events (participants affected / at risk) | 2/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PET Imaging With 89Zr-DFO-Trastuzumab (N=36)
Diarrhea (Gastrointestinal disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PET Imaging With 89Zr-DFO-Trastuzumab (N=36)
Chills (General disorders) | 1
Fever (General disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-30): https://cdn.clinicaltrials.gov/large-docs/96/NCT02023996/Prot_SAP_000.pdf